CLINICAL TRIAL: NCT06316830
Title: Randomized Clinical Trial of a 16 mg vs. 24 mg Maintenance Daily Dose of Buprenorphine to Increase Retention in Treatment Among People With Opioid Use Disorder
Brief Title: Identifying Optimal Buprenorphine Dosing for Opioid Use Disorder Treatment and Prevention of Overdose
Acronym: Optimal Bup
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Francesca Beaudoin, Professor of Epidemiology and Emergency Medicine, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000075
Record Dates: First submitted 2024-03-06; First posted 2024-03-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Maintenance Daily Dose (24mg) (Experimental): The experimental intervention is a high daily maintenance dose of buprenorphine (24 mg) plus any usual clinical care the participant receives at the clinic. This high daily dose is the upper limit of the FDA-approved dose range and was selected based on preclinical studies, clinician anecdotes, case reports, and retrospective analyses suggesting improved effectiveness of higher buprenorphine doses among patients with a history of fentanyl use. Underlying pharmacodynamic principles support that the 24 mg daily dose of buprenorphine is likely to be well-tolerated, safe, and better control cravings among people with a history of fentanyl use.
  Interventions: Drug: Buprenorphine
- Standard Maintenance Daily Dose (16mg) (Active Comparator): The control intervention is the FDA-recommended target daily maintenance dose of buprenorphine (16 mg) plus any usual clinical care the participant receives at the clinic.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine in a highly effective treatment for opioid use disorder (OUD). Buprenorphine dose guidelines for OUD treatment were determined by clinical trials conducted in populations with a history of heroin use. However, fentanyl is changing the calculation of treatment, and optimal buprenorphine dosing for people who use fentanyl is unknown.

SUMMARY:
The investigators aim to test the effectiveness of a high maintenance daily dose of buprenorphine (24 mg) for improving outcomes among patients who used fentanyl compared to the standard daily dose (16 mg).

The main question it aims to answer is: will patients who are randomly assigned to the high 24 mg maintenance dose, as compared to patients randomly assigned to the standard 16 mg maintenance dose, have improved retention in buprenorphine treatment (primary outcome), improved treatment response based on use of non-prescribed opioids (secondary outcome), decreased opioid cravings (secondary outcome), and decreased risk of fatal and non-fatal opioid overdose (exploratory outcome).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 years-old or older
* Identified by the treating physician as having moderate to severe opioid use disorder (OUD)
* Initiating or continuing buprenorphine for treatment of opioid use disorder
* History of fentanyl use (confirmed by fentanyl positive urine drug screen (UDS) at intake OR if on buprenorphine maintenance treatment fentanyl plus a positive UDS within the last month OR self- reported ongoing fentanyl use during treatment)

Exclusion Criteria:

* Previous enrollment in the trial
* Incarcerated or in police custody*
* Pregnant
* Live outside of Rhode Island (RI)
* Unable to provide informed consent
* Allergy to Buprenorphine
* Concomitant medication use deemed to present potential for serious medication interaction by the treating clinician *Participants that become incarcerated/or in police custody during the study will be withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Engagement | six months post-randomization
  The primary outcome is the percentage of participants retained in buprenorphine treatment. Participants will be classified as retained in buprenorphine treatment at six months post- randomization if (1) the study site data indicate that they remained engaged in treatment or (2) the PDMP suggest that they continued treatment elsewhere and have not had a gap of more than 27 days in medication on-hand based on fill dates and days' supply.

SECONDARY OUTCOMES:
Control of Opioid Cravings | six months post-randomization
  Measured using patient reported outcomes via the Opioid Craving Scale, a reliable, validated scale for people with opioid use disorder. The scale consists of three questions related to opioid cravings rated on a scale of 1-10 with 1 being not at all and 10 being extremely. A higher score denotes increased opioid cravings.
Treatment response based on use of non-prescribed opioids | six months post-randomization
  Non-prescribed fentanyl and other opioid use will be assessed via urine drug screens including fentanyl (UDS) and self-report. UDS will be assessed monthly for six months after study enrollment. Self-reported will be assessed at 1, 3, and 6 months via a Time Line Followback (TLFB) assessing ongoing non-prescribed opioid/fentanyl over the preceding two weeks. Based on UDS and self-reported data, participants will be classified as treatment responders if they have (1) no evidence (negative UDS and negative self-report) of non-prescribed opioid use at ≥1 assessment in months 1 to 3 AND (2) no evidence of non-prescribed opioid use at ≥2 assessments in months 4 to 6.

OTHER OUTCOMES:
Rate of Non-fatal or Fatal Opioid Overdose | twelve months post-randomization
  Non-fatal and fatal opioid overdoses will be assessed using statewide data from the Rhode Island Department of Health, including the Emergency Medical Services (EMS) Information System, Opioid Overdose Reporting System (OORS), and Office of the State Medical Examiners (OSME). All of these systems report non-fatal or fatal opioid overdoses which investigators will aggregate to arrive at the rate of non-fatal or fatal opioid overdoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon request in accordance with the policies and procedures of the Brown University and Rhode Island Department of Health Institutional Review Boards and collaborating state and local institutions
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be made available upon request

REFERENCES:
- [Background] Chambers LC, Hallowell BD, Zullo AR, Paiva TJ, Berk J, Gaither R, Hampson AJ, Beaudoin FL, Wightman RS. Buprenorphine Dose and Time to Discontinuation Among Patients With Opioid Use Disorder in the Era of Fentanyl. JAMA Netw Open. 2023 Sep 5;6(9):e2334540. doi: 10.1001/jamanetworkopen.2023.34540. PMID 37721749
- [Derived] Armeni K, Chambers LC, Peachey A, Berk J, Langdon KJ, Peterson L, Beaudoin FL, Wightman RS. Randomised clinical trial of a 16 mg vs 24 mg maintenance daily dose of buprenorphine to increase retention in treatment among people with an opioid use disorder in Rhode Island: study protocol paper. BMJ Open. 2024 Nov 9;14(11):e085888. doi: 10.1136/bmjopen-2024-085888. PMID 39521460